CLINICAL TRIAL: NCT03780894
Title: Transfusion of Red Blood Cells (RBC), Tranexamic Acid (TXA) and Fibrinogen Concentrate (FC) for Severe Trauma Hemorrhage at Pre-hospital Phase of Care. A Pilot Trial.
Brief Title: Transfusion of Red Blood Cells, Tranexamic Acid and Fibrinogen Concentrate for Severe Trauma Hemorrhage at Pre-hospital Phase of Care.
Acronym: PRETIC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRETIC
Record Dates: First submitted 2018-12-12; First posted 2018-12-19 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Polytrauma; Traumatic Hemorrhage
Keywords: Polytrauma; Red blood cells transfusion; Acute traumatic hemorrhage
MeSH Terms: conditions — Multiple Trauma | interventions — Fibrinogen; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Single-center, non-randomized, open-label, two-arms, controlled pilot clinical trial.
  The experimental and control arms will be determined according to the SEM units with RBC, TXA and FC administration capacity (i.e. helicopter unit, rapid intervention ambulance or advanced life support ambulance). The emergency SEM units are activated according current protocols based on distance, severity and weather conditions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental treatment (Experimental): The active treatment consists of intravenous injection of 2g of fibrinogen concentrate, 1g of tranexamic acid, 2 red bood cells concentrate O Rh(D) negative (Banc de Sang i Teixits, Barcelona, Spain), and crystalloids at pre-hospital phase of care.
  Interventions: Drug: Fibrinogen Concentrate (Human) 1 MG [RiaSTAP]; Biological: Red blood cells concentrate; Drug: Tranexamic Acid
- Standard treatment (Active Comparator): Patients in the control arm will be treated according the existing protocols based on crystalloids and tranexamic acid administration.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Fibrinogen Concentrate (Human) 1 MG [RiaSTAP] — Administration of 2 mg of FC together with RBC and TXA
  Arms: Experimental treatment
Biological: Red blood cells concentrate — Administration of 2 red blood cells concentrates together with FC and TXA
  Arms: Experimental treatment
Drug: Tranexamic Acid — Administration of 1g of TXA together with FC and RBC

SUMMARY:
This is a single-center, not-randomized, open-label, controlled pilot clinical trial. This study compares presence of Trauma Induced Coagulopathy (TIC) and acute traumatic hemorrhage treatment at pre-hospital phase of care with red blood cells (RBC), Tranexamic acid (TXA) and Fibrinogen Concentrate (FC) with the current treatment based on the administration of Crystalloids and TXA.

DETAILED DESCRIPTION:
A pilot, non-randomized, open-label study of two intervention arms and controlled with the standard treatment in which 60 patients affected with acute hemorrhage due to severe trauma will enter the study with the main objective of evaluating the feasibility and the efficacy of early treatment during the pre-hospital care phase with packed red blood cells, fibrinogen concentrate and tranexamic acid (experimental arm) compared to the standard treatment based on crystalloids administration and tranexamic acid (control arm). The secondary objectives are to evaluate the safety and clinical evolution of the patients. Prior to the administration of the treatment, 2 blood samples will be extracted in both groups in order to compare the coagulation status and to be able to perform the pre-transfusion tests. On arrival at the hospital, another sample will be taken to compare changes in coagulation after the administration of the experimental or standard treatment and also between both groups. The assessment of the coagulation status will be made using the values provided by the viscoelastic test (TEG6s). The experimental and standard treatment will be administered endovenously. After treatment, patients will be evaluated up to 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years AND
* Patients with severe trauma categorized as priority 0 or 1 according to the CatSalut Polytrauma Code (PPT) AND
* Evidence of bleeding or a high bleeding suspicion according to physician judgment OR
* Predicted to need transfusion according to TICCS score ≥10

Exclusion Criteria:

* Moribund patient with devastating injuries and expected to die within 1-hour OR
* Known objection to blood components transfusion OR
* Known acquired or congenital coagulopathies not related to the actual trauma OR
* Known anticoagulant treatment (vitamin K antagonist, dabigatran, rivaroxaban, apixaban) OR
* Known Pregnancy OR
* Severe isolated traumatic brain injury OR
* Hemorrhage not related to the actual trauma

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2021-01-11 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
TEG6s(R) parameters for Trauma Induced Coagulopathy (TIC) | Basal (at the crash site)
  TEG6s(R) parameters that define TIC
TEG6s(R) parameters for Trauma Induced Coagulopathy (TIC) | Basal (at the hospital arrival)
  TEG6s(R) parameters that define TIC
All-cause mortality | 1 hour post hospital admission
  Mortality for any cause
All-cause mortality | 6 hours post hospital admission
  Mortality for any cause
All-cause mortality | 24 hours post hospital admission
  Mortality for any cause
Accountability | 30 days
  Red bood cells concentrate accountability
Temperature storage conditions of the red blood cells concentrate | 24 hours
  Red bood cells concentrate out of temperature range for storage

SECONDARY OUTCOMES:
All-cause mortality | 48 hours post hospital admission
  Mortality for any cause
All-cause mortality | 30 days post hospital admission
  Mortality for any cause
Adverse Events | 30 days post hospital admission (or previously at hospital discharge)
  Treatment emergent adverse events
Thromboembolism events | 30 days
  Thromboembolism events
Crystalloid fluid requirements | 1 hour (from the crash site to the hospital admission)
  Volume of crystalloids required
Crystalloid fluid requirements | 30 days post hospital admission (or previously at hospital discharge)
  Volume of crystalloids required
Transfusion requirements | 24 hours (or previously at discharge of the emergency room)
  Transfusion requirements of RBC, platelets and plasma
Transfusion requirements | 30 days post hospital admission (or previously at hospital discharge)
  Transfusion requirements of RBC, platelets and plasma
Water balance | 24 hours of admission at the ICU
  Water balance at the Intensive Care Unit (ICU)
Water balance | 72 hours of admission at the ICU
  Water balance at the Intensive Care Unit (ICU)
Ventilator-free days | 30 days
  Ventilator-free days at the ICU

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Blood and Tissue Bank of Catalonia — http://www.bancsang.net
- See also: HOspital Universitari Dr. Trueta (Girona, Spain) — http://icsgirona.cat